CLINICAL TRIAL: NCT04140929
Title: Oral Health Improvement for Nursing Home Residents Through Delegated Remotivation and Reinstruction - a Cluster-randomized Controlled Trial
Brief Title: Oral Health Improvement for Nursing Home Residents Through Delegated Remotivation and Reinstruction
Acronym: MundZaRR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Jena University Hospital (Other); Martin-Luther-Universität Halle-Wittenberg (Other); University of Applied Sciences, Cologne, Germany (Unknown); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katrin Hertrampf, Principle Investigator, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01VSF18021
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2023-12

CONDITIONS: Oral Health; Oral-health Associated Quality of Life
Keywords: nursing homes; oral hygiene; quality of life; health services research

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): In the intervention group, a range of clinical parameters are recorded and the dentists prepares an individual oral hygiene and care recommendation, based on the Oral Health Tool Box. The Box is also used for instructing the dental assistants and the nursing staff for each patient individually. It is then determined when and how the dental assistants re-evaluates the oral hygiene and care process and reinstructs and remotivates the nursing staff. If the examination reveals a need for dental treatment (possibly requiring referral and transport), this will be communicated to the nursing staff. The dental assistant will further receive a training in communication, enabling them in reinstruction and remotivation. Dentists and dental assistants will further receive a training in geriatric dentistry by the State Commissioner of the German Society for Geriatric Dentistry.
  Interventions: Other: Oral Health Tool Box
- Control group (No Intervention): In the control group, the residents receive care as usual. This includes the recording of the same parameters are recorded as in intervention group, a standardized form is filled out and handed over to the nursing staff. As in the case of Intervention group, the nursing staff is informed in the event of a need for treatment. No further measures are applied.

INTERVENTIONS:
Other: Oral Health Tool Box — Please see, description of the intervention group
  Arms: Intervention group

SUMMARY:
Based on the poor situation of residents in German nursing homes with regard to oral health, a cluster-randomized Trial will be carried out in Rhineland-Palatindate, Germany. Dentists investigated residents to identify dental or oral hygiene problems. In the invention group, dentists' recommendations will be reinstructed to the nursing staff by dental assistance.

DETAILED DESCRIPTION:
Introduction: Oral health and oral-health-associated quality-of-life (OHrQL) of residents in German nursing homes are poor. The investigators will develop an evidence-based catalogue of interventions applicable and sustainable ("Oral Health Tool Box"). Based on this, care-accompanying reinstruction and remotivation of nursing staff by dental assistants (DA) will be provided. The investigators hypothesize such complex intervention to significantly improve OHrQL, and daily oral hygiene/care behaviour and its cost-effectiveness.

Methods and analysis: Based on the findings of a rapid systematic review, possible intervention components will be systematized and assessed for their effectiveness. Mixed methods will be used to identify barriers and enablers of oral hygiene and care in German long-term residential care (LRC), and these will be linked with the intervention components using the Theoretical Domains Framework and the Behavior Change Wheel, the result being an "Oral Health Tool Box". A two-arm cluster, randomized-controlled-trial (ratio of 1:1 via block randomization) will be performed in nursing homes in Rhineland-Palatinate, Germany, including residents with moderate to severe care dependency. Each nursing home represents a cluster. Based on a feasibility study, considering clustering and possible attrition, the investigators aim at recruiting 618 residents of 18 cluster. In the intervention group, dentists will identify the specific problems of each resident, and assign one or more intervention components from the box. During follow-up, nursing staff will be reinstructed and remotivated by dental assistants in how to deliver the intervention components in individual intervals. In the control group residents will receive care as usual. The primary outcome, OHrQL, will be measured using the German version of the General Oral Health Assessment Index (GOHAI). Secondary outcomes include pain condition, general health-related quality-of-life, caries increment, oral/prothetic hygiene and gingival status, incidence of dental emergencies and hospitalizations, and cost-utility/effectiveness. The endpoints will be measured at baseline and after 12 months. For the primary outcome, a mixed-linear model will be used within an intention-to-treat analysis. A process evaluation using mixed methods will be conducted alongside the trial.

Due to the pandemic, the number of cases could not be reached despite outstanding commitment in recruitment. An application was made to the funding agency to adapt the project plan.

ELIGIBILITY:
Inclusion Criteria:

* Nursing homes without an existing dental cooperation agreement. Eligible are residents with a degree of care dependency of 3 to 5 (moderate to severe) as rated by an expert rater of the German statutory health insurance.

Exclusion Criteria:

* lack of consent (of the home management and/or the residents or their proxies or legal guardians) and residents in respite carer

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
General Oral Health Assessment Index (GOHAI) | 12 months
  The GOHAI is an established instrument for measuring oral health-related quality of life (OHRQoL) in older people. It comprises twelve items in four domains (functional limitations, pain/discomfort, psychological aspects, behavioral aspects), which are recorded ordinally scaled from 0 (never true) to 5 (always true).

SECONDARY OUTCOMES:
Pain scale | 12 months
  Measurement of actual pain by scale (1-10), 1 -least pain, 10-most pain
European Group Quality of life-5 Dimenions-5 Levels (EQ-5D-5L) | 12 months
  Health-related quality of life
Decayed-Missing-Filled-Teeth (DMFT) | 12 months
  Caries experience/tooth loss, measured with Decayed-Missing-Filled Teeth,and root caries lesions
Geriatric Debris Index (GDI-S) | 12 months
  Oral hygiene status
Periodonal Sulcus Index (PSI) | 12 months
  gingival inflammation
Denture Hygiene Index | 12 months
  Prosthetic hygiene
Health economic analysis | 12 months
  Incidence of dental-associated emergencies and hospitalisations. Nursing,dental and inpatient treatment costs

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Schleswig-Holstein, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
After completion of the whole study, the results will be published

REFERENCES:
- [Derived] Nordblom NF, Hertrampf K, Habig S, Gabelmann S, Schlattmann P, Orawa H, Meyer G, Gassmann G, Abraham J, Wobst LM, Schwendicke F. Cost-effectiveness-analysis of oral health remotivation and reinstruction in nursing homes in a cluster-randomized controlled trial. J Dent. 2025 Feb;153:105520. doi: 10.1016/j.jdent.2024.105520. Epub 2024 Dec 13. PMID 39673909
- [Derived] Hertrampf K, Schlattmann P, Meyer G, Gassmann G, Abraham J, Hammen V, Schwendicke F. Oral health improvement for nursing home residents through delegated remotivation and reinstruction (MundZaRR Study): study protocol of a cluster-randomised controlled trial. BMJ Open. 2020 Sep 25;10(9):e035999. doi: 10.1136/bmjopen-2019-035999. PMID 32978183